CLINICAL TRIAL: NCT03795142
Title: A Phase I Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BGB149 Following Single Dose Administration in Healthy Subjects
Brief Title: A First-time-in-human Study of BGB149
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: BerGenBio ASA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Screening
Other Study IDs: BGB149-101
Record Dates: First submitted 2018-11-23; First posted 2019-01-07 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The clinical study will be performed in a double-blinded manner for all cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single intravenous dose; BGB149 (Experimental): A single intravenous dose of BGB 149 or matched placebo will be administered on day 1 ascending doses will be administered in cohorts of 6 (randomised 4:2, active: placebo) at a planned four dose levels (maximum of six dose levels to be investigated under initial approved protocol) A sentinel cohort of 2 volunteers will randomly receive (1:1) either experimental or matched placebo infusion
  Interventions: Biological: BGB149
- single intravenous dose; placebo (Placebo Comparator): A single intravenous dose of BGB 149 or matched placebo will be administered on day 1 ascending doses will be administered in cohorts of 6 (randomised 4:2, active: placebo) at a planned four dose levels (maximum of six dose levels to be investigated under initial approved protocol) A sentinel cohort of 2 volunteers will randomly receive (1:1) either experimental or matched placebo infusion
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BGB149 — Single Ascending Dose
  Arms: single intravenous dose; BGB149
Biological: Placebo — Matching placebo
  Arms: single intravenous dose; placebo

SUMMARY:
This clinical trial is a Phase I, first-in-human. The study is designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of BGB149 after single IV doses in healthy male and female subjects. Multiple dose levels will be explored.

ELIGIBILITY:
Inclusion Criteria:

* The subject voluntarily agrees to participate in this study and signs an Independent Ethics Committee approved informed consent form prior to performing any of the screening procedures.
* Healthy male and female subjects, between 18 to 55 years of age, inclusive, at the screening visit.
* If male, Must agree to use appropriate double-barrier contraception and to refrain from donating sperm from the time of dosing until 3 months after dosing.
* If female, Must be of non-childbearing potential (surgically sterile [hysterectomy or bilateral tubal ligation] or postmenopausal ≥ 1 year with follicle stimulating hormone > 40 IU/L).
* Body mass index between 18.0 and 30.0 kg/m2, inclusive, at the screening visit with a weight of at least 50kg.
* Non-smoker, defined as a subject who has not smoked previously and/or who has discontinued smoking or the use of nicotine/nicotine-containing products (including snuff and similar products) at least 3 months before the screening visit.
* Subjects are in good health, as determined by medical history, physical examination, vital signs assessment, resting 12-lead ECG and clinical laboratory evaluations within normal reference ranges or outside of normal reference ranges considered not clinically relevant by the Principal Investigator or designee.
* Subject must have suitable veins for cannulation and/or repeated venipuncture.

Exclusion Criteria:

* Female subjects of childbearing potential, or breastfeeding, or have a positive serum pregnancy test at the screening visit or a positive urine pregnancy test on admission.
* A positive urine cotinine result (>500ng/mL) at the screening visit or on admission.
* Subjects who have ongoing or significant history of alcoholism or drug/chemical abuse in the past 5years, as determined by the Principal Investigator or designee.
* Subjects who have positive urine drugs of abuse screen at the screening visit or on admission, or a positive urine alcohol test at the screening visit or on admission.
* Subjects who are unwilling to avoid the use of alcohol within 48 hours before any study visit and while confined to the study center.
* Subjects who are unwilling to abstain from heavy physical training from 7 days before first dosing until the final follow-up visit.
* Subjects who have used the following: Any prescribed medication within 14 days prior to planned time of dosing. Non-prescription or over-the-counter medication, herbal and dietary supplements such as St John's Wort, vitamins and minerals that could affect the outcome of the study within 1 week prior to planned time of dosing. Live attenuated vaccines and systemic corticosteroids within 3 months prior to planned time of dosing.
* Subjects who have donated blood in the 3 months prior to the screening visit, plasma in the 7 days prior to the screening visit or platelets in the 6 weeks prior to the screening visit.
* Subjects who have a history of significant drug allergy (e.g., anaphylaxis) or any clinically significant allergic condition (excluding non-active hay fever), as determined by the Principal Investigator or designee.
* Subjects who have had a clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of dosing, as determined by the Principal Investigator or designee.
* Subjects with history of gastrointestinal bleeding or ulceration or perforation; history of Crohn's disease or any other inflammatory disorder of the gastrointestinal tract.
* Subjects with history of bone marrow transplant, with or without graft versus host disease.
* Subjects who have pulse, blood pressure, respiratory rate or oral body temperature values outside the normal ranges at the screening visit or on admission that is, in the opinion of the Principal Investigator or designee, clinically relevant and increases the risk of participating in the study.
* Results of alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) and/or total bilirubin (TBL) above the upper limit of normal (ULN), as confirmed by subsequent repeat assessment, at the screening visit and on admission.
* A positive serology test for hepatitis A virus IgM antibodies (anti-HAV IgM), hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, or antibodies to human immunodeficiency virus (HIV) Type 1 and/or Type 2 at the screening visit.
* Subjects who are still participating in another clinical study or received last study drug dose in a clinical study within 3 months or 5 half-lives, prior to dosing in this study, whichever is longer.
* Employees of the Sponsor or the contract research organization (CRO), with direct involvement in the proposed study or other studies under the direction of the Principal Investigator or the CRO, as well as close relatives of the employees.
* Subjects who are unlikely to comply with the protocol requirements, instructions and study related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits and improbability of completing the clinical study.
* Vulnerable subjects defined as individuals whose willingness to volunteer in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate (e.g., persons in detention, minors and those incapable of giving consent).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent clinical adverse events (AE) following single intravenous (IV) administration of BGB149 or matched placebo | 85 days
  Number of healthy volunteers experiencing adverse events (AE) AE categorized by grading for severity according to the Common Terminology Criteria for Adverse Events (CTCAE version 5.0).
Frequency of treatment-emergent laboratory abnormalities following single intravenous (IV) administration of BGB149 or matched placebo | 85 days
  Number of healthy volunteers experiencing clinically significant abnormalities of clinical laboratory tests (hematology, coagulation, clinical chemistry and urinalysis); categorized by grading for severity according to the CTCAE version 5.0.

SECONDARY OUTCOMES:
Pharmacokinetic Parameters: BGB149 Cmax following single intravenous (IV) administration of BGB149 or matched placebo | 85 days
  Cmax: measured maximum BGB149 concentration, determined directly from the concentration-time profile.
Pharmacokinetic Parameters: BGB149 Tmax following single intravenous (IV) administration of BGB149 or matched placebo | 85 days
  Tmax: Time of maximum BGB149 concentration determined directly from the concentration-time profile.
Pharmacokinetic Parameters: BGB149 AUC(0-last), following single intravenous (IV) administration of BGB149 or matched placebo | up to 85 days
  Area under the concentration-time curve from pre-dose (time 0) to the time of the last quantifiable concentration calculated using the linear-log trapezoidal rule.
Pharmacokinetic Parameters: BGB149 AUC(0-infinity) following single intravenous (IV) administration of BGB149 or matched placebo | 85 days
  Area under the concentration-time curve from pre-dose (time 0) extrapolated to infinite time (AUClast + Clast/Lambda[z]) calculated using the linear-log trapezoidal rule.
Pharmacokinetic Parameters: BGB149 terminal elimination rate constant λz, following single intravenous (IV) administration of BGB149 or matched placebo | 85 days
  λz: The terminal elimination rate constant determined by selection of at least three data points on the terminal phase of the concentration-time curve.
Pharmacokinetic Parameters: BGB149 t½: Terminal elimination half-life, following single intravenous (IV) administration of BGB149 or matched placebo | 85 days
  t½: Terminal elimination half-life calculated as: ln2/λz
Pharmacokinetic Parameters: BGB149 total body clearance (CL) following single intravenous (IV) administration of BGB149 or matched placebo | 85 days
  CL: Total body clearance
Immunogenicity indicators: anti-drug antibodies [ADA] | 85 days
  Immunogenicity - Detection and titre of anti-drug antibodies [ADA], determined using a validated assay.
Immunogenicity indicators: neutralizing antibodies [NAb] | 85 days
  Immunogenicity - Detection and titre of neutralizing antibodies [NAb], determined using a validated assay (titres and NAb analyses performed when ADA screening is positive
Pharmacodynamics: detection of soluble Axl protein in circulation | 85 days
  PD - Concentration of soluble Axl measured in serum after dosing, determined using a validated assay.

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, MD, Principal Investigator — Parexel
Locations (1):
- Parexel Northwick Park, London, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No